CLINICAL TRIAL: NCT01845779
Title: Evaluation of Immune Response Against Human Papillomavirus (HPV)in Patients With Metastatic Cancer of the Anal Canal
Acronym: Epitopes-HPV01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Epitope-HPV01
Record Dates: First submitted 2013-04-15; First posted 2013-05-03 (Estimated); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Metastatic Anal Canal Cancer; Human Papillomavirus
MeSH Terms: conditions — Anal Canal Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- patients in complete response (Experimental)
  Interventions: Drug: DCF regimen

INTERVENTIONS:
Drug: DCF regimen

SUMMARY:
Complete response is a rare event in metastatic anal cancer in the case of unresectable recurrence after radiochemotherapy.

In the University Hospital Center of Besançon, 8 patients with metastatic anal cancer were treated between 2005 and 2008 by 6 cycles of chemotherapy including taxane: DCF (Docetaxel, Cisplatin and 5-Fluorouracil.

In more than 90% of cases, anal cancers are related to Human Papilloma Virus (HPV) infection, that is the case of this patients for which HPV16 (human papillomavirus type 16) genotype was identified within the tumor samples.

The hypothesis is that an anti-HPV response immune could be generated by chemotherapy with DCF and contributed to the elimination of the tumour cells and to the increase of complete responses. The aim to this study is to analyze immune response against HPV in this patients in complete response.

ELIGIBILITY:
Inclusion Criteria:

* ECOG performance status ≤ 1
* patient with metastatic anal cancer HPV+
* presence of a measurable target lesion according to radiological criteria (Recist V1.1)
* patient with more than 12 months of complete remission of metastatic anal cancer according to radiological criteria (Recist V1.1)after treatment by DCF regimen (Docetaxel, Cisplatin and 5-Fluorouracil)

Exclusion Criteria:

* pregnancy or lactation
* patient with any medical or psychiatric condition or disease which would make the patient inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
presence and characterization of anti-HPV immune responses in patients in complete remission | 3 months after sample

SECONDARY OUTCOMES:
global survival | from date to initiation of chemotherapy until the date of death for any cause assessed up to 100 months
progression free survival | from date to initiation of chemotherapy until the date of first documented progression, assessed up to 60 months

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Oncology - University Hospital of Besançon, Besançon, France